CLINICAL TRIAL: NCT06860152
Title: O15-PET Imaging of Cochlear Implant Speech in Noise Processing
Brief Title: Cochlear Implant Speech in Noise Processing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phillip Gander (Other)
Responsible Party: Sponsor-Investigator, Phillip Gander, Research Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202403834
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Hearing Loss, Adult-Onset; Speech Intelligibility; Hearing Loss, Extreme
MeSH Terms: conditions — Hearing Loss; Speech Intelligibility; Deafness | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cochlear implant (Experimental): Experienced (greater than 1 year) cochlear implant recipients
  Interventions: Device: Cochlear implant
- Age-typical hearing control (No Intervention): Age-matched, age-typical (normal) hearing control participants

INTERVENTIONS:
Device: Cochlear implant — Cochlear implant
  Arms: Cochlear implant

SUMMARY:
The study will help us in understanding the neural mechanisms by which listeners with a cochlear implant detect speech in noisy environments.

DETAILED DESCRIPTION:
Despite the success of a cochlear implant (CI) for providing or improving hearing ability for people with severe hearing loss, everyday conversations in background noise are still the main clinical complaint. The goal of this study is to understand the neural mechanisms by which listeners with a CI detect speech in noisy environments, and to understand how these mechanisms differ across a variety of CI listeners, in order to determine what variables are most relevant for predicting successful outcome. Therefore the purpose of PET neuroimaging in this study is to find the brain regions that relate to speech in noise effort using PET during auditory stimulation on a single session across a variety of CI users with different device configurations. An age-matched typical hearing control group provides a baseline for comparison. PET neuroimaging will be performed using a radioactive form of water, O-15 (an investigational agent), that will be injected into the body to examine brain blood flow using a PET/CT scanner.

ELIGIBILITY:
Cochlear Implant subjects (enrollment is planned at N=120) - Inclusion criteria:

1. Between 18 and 99 years of age.
2. Have a cochlear implant activated for more than one year.
3. Eligible for research under the Iowa Cochlear Implant Project VIII.
4. Ability to understand and willingness to sign a written informed consent document.
5. Severe hearing loss after age 16.

Normal Hearing subjects (enrollment is planned at N=30) - Inclusion criteria:

1. Between 18 and 99 years of age.
2. Have age typical hearing.
3. Eligible for research under the Iowa Cochlear Implant Project VIII.
4. Ability to understand and willingness to sign a written informed consent document.

Exclusion criteria (all groups):

1. Medical history includes seizure disorder, head injury, neurologic, metabolic, cardiovascular disease, or previous cerebrovascular event (unless approved by PI).
2. Female self-reporting pregnancy. A urine pregnancy test will be performed prior to injection of the radiopharmaceutical.
3. Currently taking medications which may affect cerebral blood flow (e.g., papaverine, ginkgo biloba, acetazolamide).
4. Uncontrolled intercurrent illness that would limit compliance with study requirements per investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
To identify the cortical bases for speech-in-noise understanding in cochlear implant users | Basline Visit
  PET imaging will be used to identify the brain regions for listeners ability to recognize speech in noise at different signal-to-noise ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip E. Gander, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No